CLINICAL TRIAL: NCT03629600
Title: A Prospective Open-label Randomized Controlled Trial Comparing Effectiveness of Aggressive Hydration Versus High-dose Rectal Indomethacin in the Prevention of Post-ERCP Pancreatitis (PEP)
Brief Title: Trial of Aggressive Hydration Versus Rectal Indomethacin for Prevention of Post-ERCP Pancreatitis
Acronym: AHRI-PEP
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Kshaunish Das, Professor, Division of Gastroenterology, SDLD, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IEC/2016/396
Record Dates: First submitted 2018-08-09; First posted 2018-08-14 (Actual); Last update posted 2018-08-16 (Actual); Status verified 2018-08

CONDITIONS: Post-ERCP Acute Pancreatitis
MeSH Terms: interventions — Ringer's Lactate

STUDY DESIGN:
Intervention Model Description: Prospective randomized open-label parallel-group non-inferiority controlled clinical trial
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aggressive Hydration (Experimental): Patients randomized to the aggressive intravenous hydration group received Lactated Ringers solution (LR) [COMPOUND SODIUM LACTATE INJECTION I.P.,INVEN PHARMACEUTICALS PVT.LTD,MP,INDIA] intravenously (IV) at 3 mL/kg/hr during the ERCP, a 20cc/kg IV bolus immediately afterward, and then at 3 mL/kg/hr for 8 hours following the procedure.
  Interventions: Drug: Lactated Ringer
- Rectal Indomethacin (Active Comparator): Patients randomised to Rectal Indomethacin were administered a suppository of 100 mg of indomethacin [Indomethacin Suppository 100 Mg B.P, GALEN PHARMACEUTICAL LTD, GUJRAT, INDIA] just after the completion of ERCP procedure.
  Interventions: Drug: Rectal Form Indometacin

INTERVENTIONS:
Drug: Lactated Ringer — High-volume Lactated Ringer Solution
  Other Names: COMPOUND SODIUM LACTATE INJECTION I.P., INVEN PHARMACEUTICALS PVT.LTD, MP, INDIA
  Arms: Aggressive Hydration
Drug: Rectal Form Indometacin — Post-ERCP rectal administration of 100 MG Indomethacin
  Other Names: INDOMETHACIN SUPPOSITORY 100 Mg B.P, GALEN PHARMACEUTICAL LTD, GUJRAT, INDIA
  Arms: Rectal Indomethacin

SUMMARY:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is a commonly performed endoscopic procedure used to treat pancreato-biliary pathology. Acute pancreatitis or post-ERCP pancreatitis (PEP), is the most common major complication of ERCP, which is reported to occur in 2-10% of patients overall (ranging from 2-4% in low risk patients up to 8-40% in high-risk patients). Hydration is a mainstay of treatment for acute pancreatitis, independent of etiology. Aggressive hydration has also been shown to decrease incidence of PEP. Rectal NSAIDs, including Indomethacin, has a proven role in prevention of PEP. Though both aggressive hydration and rectal indomethacin are efficacious in preventing PEP, there is no head to head trial comparing the efficacy of these two therapeutic modalities. Thus, the aim is to determine whether aggressive intravenous peri-procedural hydration or high dose rectal indomethacin immediately after ERCP decrease the incidence of PEP. The investigator's hypothesis is that prophylactic treatment with aggressive intravenous hydration is not inferior to rectal indomethacin in preventing PEP.

DETAILED DESCRIPTION:
Endoscopic Retrograde Cholangiopancreatography (ERCP) is a commonly performed endoscopic procedure used to treat pancreato-biliary pathology. Acute pancreatitis is the most common major complication of (ERCP)[1] which is reported to occur in 2-10% of patients overall (ranging from 2-4% in low risk patients up to 8-40% in high-risk patients) [1, 2]. The wide range of reported incidence of post-ERCP pancreatitis over risk groups in observational studies prompted a 2014 systematic review including 108 RCTs that covered 13 296 patients[3]. The overall incidence of post-ERCP pancreatitis was 9.7%, of which 8.6% of cases were mildly severe, 3.9% were moderate,and 0.8% were severe. The incidence of all-severity post-ERCP pancreatitis in high-risk patients was 14.7%. This study also found, however, that the incidence of severe post-ERCP pancreatitis (0.5% of all ERCPs performed) did not differ between patients in a high-risk subgroup and non-risk-stratified RCTs (0.8% vs. 0.4%, respectively), perhaps due to heterogeneity between the RCTs regarding the risk assessment of patients

The generally accepted criteria for the diagnosis of post-ERCP pancreatitis were proposed in 1991 during a consensus workshop. These criteria include new onset of pancreatic-type abdominal pain associated with at least a threefold increase in serum amylase or lipase occurring within 24 h after ERCP, and the pain symptoms need to be sufficiently severe to require admission to the hospital or to extend the length of stay of patients who are already hospitalized [3].

Hydration is a mainstay of treatment for acute pancreatitis, independent of etiology[4]. Experiments in animal models demonstrate that pancreatic microvascular hypoperfusion leads to necrosis[5]. Clinical studies of fluid resuscitation in patients with acute pancreatitis suggest that hemoconcentration and decreased systemic perfusion are associated with increased risk of pancreas necrosis and unfavorable outcome [6]. Hydration has also been shown to decrease incidence of PEP.

Besides Hydration, rectal NSAIDS, including Indomethacin, has role in prevention of post ERCP Acute pancreatitis. Though both aggressive hydration and rectal indomethacin are efficacious in preventing Post ERCP pancreatitis there is no head to head trial comparing the efficacy of these two therapeutic modality.

To determine whether aggressive intravenous peri-procedural hydration or high dose rectal indomethacin immediately after ERCP decrease the incidence of post ERCP pancreatitis.

The investigator's hypothesis is that prophylactic treatment with aggressive intravenous hydration is not inferior to rectal indomethacin in protecting against Post ERCP pancreatitis .

ELIGIBILITY:
Inclusion Criteria:

* All patients aged 18 to 70 years undegoingt ERCP for the first time
* Patients undergoing ERCP for standard clinical indications

Exclusion Criteria:

* Ongoing acute pancreatitis
* Known chronic calcific pancreatitis
* Pancreatic head mass
* Any malignancy
* Standard contraindications to ERCP
* Unwillingness or inability to consent for the study
* Ongoing hypotension including those with sepsis
* Cardiac insufficiency (CI, >NYHA Class II heart failure)
* Renal insufficiency (RI, creatinine clearance <40mL/min)
* Severe liver dysfunction (albumin < 3mg/dL)
* Respiratory insufficiency (defined as oxygen saturation < 90%)
* Greater than 70 years of age
* Pregnancy
* Breastfeeding mother
* Allergy/hypersensitivity to aspirin or NSAIDs
* Received NSAIDs in prior 7 days (aspirin 325mg or less ok)
* Active or recurrent (within 4 weeks) gastrointestinal hemorrhage
* Hyponatremia (Na+ levels < 135mEq/L))
* Hypernatremia (Na+ levels > 150mEq/L) will be excluded.
* Edema or anasarca
* Ascites
* Procedure performed on major papilla/ventral pancreatic duct in patient with pancreas divisum (dorsal duct not attempted on injected)
* ERCP for biliary stent removal or exchange without anticipated pancreatogram
* Subject with prior biliary sphincterotomy now scheduled for repeat biliary therapy without anticipated pancreatogram
* Anticipated inability to follow protocol

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 352 (Actual)
Dates: Start 2017-10-15 (Actual); Primary Completion 2018-02-15 (Actual); Study Completion 2018-05-31 (Actual)

PRIMARY OUTCOMES:
Post-ERCP Acute Pancreatitis | 24 hours
  The primary endpoint is development of post-ERCP pancreatitis (PEP, a categorical variable) which will be defined as presence of increased abdominal pain and a serum amylase level three times the upper limit of normal (3xULN). Increased pain will be defined as an increase in the visual analog pain score compared to the value immediately prior to ERCP

SECONDARY OUTCOMES:
Clinical volume overload | 24 hours
  Clinical volume overload was defined by physical findings of lower extremity edema and pulmonary rales.
Serum Amylase three times the upper limit of normal | 8 hours
  Serum amylase three times the upper limit of normal is a secondary outcome measure. (Measured with α-Amylase KIT by direct substrate method; BEACON DIAGNOSTICS PVT LTD, INDIA)
Post-ERCP pain abdomen: VAS | 24 hours
  Patients admitted with pain abdomen after ERCP for less than 24 hrs. Increased abdominal pain is defined as an increase in abdominal pain based on the visual analogue score following the ERCP compared to the score immediately prior to the ERCP.

OTHER OUTCOMES:
Death | 7 days
  Death within 7 days after performing ERCP

CONTACTS AND LOCATIONS:
Overall Officials: Kshaunish Das, MD, DM, Principal Investigator — Professor, Division of Gastroenterology, SDLD, IPGMER
Locations (1):
- IPGIMER, Kolkata, West Bengal, India

IPD SHARING:
Plan to Share IPD: Undecided
Baseline data, outcomes

REFERENCES:
- [Derived] Guha P, Patra PS, Misra D, Ahammed SM, Sarkar R, Dhali GK, Ray S, Das K. An Open-Label Randomized Controlled Trial Comparing Effectiveness of Aggressive Hydration Versus High-dose Rectal Indomethacin in the Prevention of Postendoscopic Retrograde Cholangiopancreatographic Pancreatitis (AHRI-PEP). J Clin Gastroenterol. 2023 May-Jun 01;57(5):524-530. doi: 10.1097/MCG.0000000000001712. Epub 2022 Apr 21. PMID 35470300